CLINICAL TRIAL: NCT06421805
Title: A Single-center, Prospective, and Observational Study on Population Characteristics, Pathological Features, and Prognostic Factors of Patients With Mediastinal Tumor: Establishing Mediastinal Tumor Database of PUMCH.
Brief Title: Establishing Prospective Mediastinal Tumor Database of PUMCH
Acronym: MTDPUMCH
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuehan Gao, Principal Investigator, Peking Union Medical College Hospital
Other Study IDs: MTDPUMCH
Record Dates: First submitted 2024-04-20; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Thymic Epithelial Tumor; Teratoma; Thymic Cyst; Retrosternal Goitre; Germ Cell Tumor; Lymphoma; Schwannoma
Keywords: mediastinal tumors; database; thymic epithelial tumor
MeSH Terms: conditions — Thymic epithelial tumor; Teratoma; Mediastinal Cyst; Goiter, Substernal; Neoplasms, Germ Cell and Embryonal; Lymphoma; Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — After obtaining informed consent from the patients, tumor tissue specimens will be stored in the sample repository of PUMCH at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- thymoma: mediastinal tumors_thymoma
- teratoma: mediastinal tumors_teratomas
- germ cell tumor: mediastinal tumors_germ cell tumors
- lymphoma: mediastinal tumor_lymphoma
- mediastinal neuroendocrine tumors (NETs): mediastinal tumor_NETs, including neuroendocrine tumours and neuroendocrine carcinomas.
- neurinoma: mediastinal tumor_neurinoma
- thymic carcinoma: mediastinal tumor_thymic carcinoma
- others: mediastinal tumors_other tumors

SUMMARY:
This study aims to prospectively document the population characteristics, imaging findings, pathological features, prognostic factors, etc., of patients with mediastinal tumors. Clinical information will be structured and processed, and it is recommended to establish a mediastinal tumors database at Peking Union Medical College Hospital. The goal is to provide support for the quality of diagnosis and treatment, clinical protocols, and medical decision-making related to mediastinal tumors.

DETAILED DESCRIPTION:
Mediastinal tumors encompass a variety of tumors originating in the mediastinum, comprising both benign and malignant tumors, those invading mediastinal structures during disease progression, or metastases from malignant tumors originating elsewhere in the body. Based on their relationship with the pericardium, mediastinal tumors can be categorized into anterior mediastinal tumors, commonly including thymomas, retrosternal goiters, teratomas, and germ cell tumors; middle mediastinal tumors, which often include bronchogenic cysts, lymphomas, malignant lymphomas, pericardial cysts, lipomas, and esophageal cysts; and posterior mediastinal tumors, where neurogenic tumors and neurofibromas are prevalent. Mediastinal tumors are relatively rare compared to other solid tumors and exhibit complex pathological types. Consequently, conducting prospective randomized controlled clinical trials is challenging, and the significant treatment disparities among different types of mediastinal tumors affect patient survival outcomes. Clinicians often have limited understanding of some complex mediastinal tumors due to the lack of quality and reliable diagnostic and treatment standards or survival data. Therefore, establishing a specialized database for mediastinal tumor research holds great practical significance for the effective development of clinical practice.

Tumor registration databases in North America and Europe have been established earlier, with wide coverage and relatively mature development. For example, the National Cancer Database (NCDB) in the United States is the largest tumor registration database globally, with over 1500 hospitals reporting tumor data to it, covering approximately 70% of newly diagnosed cancer cases. The Surveillance, Epidemiology, and End Results (SEER) database is a public health database based on tumor populations in some states and counties in the United States (17 regional registration centers). It has been registering data since 1973, covering tumor monitoring, epidemiology, and prognosis information. Both databases have high coverage and reasonable registration and verification systems, providing a wealth of high-level evidence for the formulation of tumor prevention and control strategies.

In China, the development in this field started relatively late. To integrate resources, deeply explore data information, and further improve the diagnosis and treatment level and patient management level of mediastinal tumors in China, it is necessary to establish a scientifically standardized specialized mediastinal tumor database.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or pathological diagnosis of mediastinal tumors;
2. Written consent is able to obtained.

Exclusion Criteria:

1. Incomplete clinicopathological information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with mediastinal tumors clinically or pathologically.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2044-12-30 (Estimated); Study Completion 2045-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of enrollment until the date of death from any cause, assessed up to 20 years
  Overall survival of patients with mediastinal tumors

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of enrollment until the date of first documented progression, assessed up to 20 years
  Progression free survival of patients with mediastinal tumors

CONTACTS AND LOCATIONS:
Overall Officials: Shanqing Li, Prof., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The research results have not been published.